CLINICAL TRIAL: NCT03817398
Title: Stopping Tyrosine Kinase Inhibitors (TKI) to Assess Treatment-Free Remission (TFR) in Pediatric Chronic Myeloid Leukemia - Chronic Phase (CML-CP)
Brief Title: Stopping Tyrosine Kinase Inhibitors in Affecting Treatment-Free Remission in Patients With Chronic Phase Chronic Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAML18P1; NCI-2018-03439 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML18P1 (Other: Children's Oncology Group); AAML18P1 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-01-02; First posted 2019-01-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia, BCR-ABL1 Positive
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Specimen Handling; Pharmaceutical Preparations; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Basic Science (stop taking TKI, biospecimen collection) (Experimental): Patients stop taking TKI medication within 10 days after enrollment. Patients undergo peripheral blood collection to monitor loss of MMR every 4 weeks in year 1, every 6 weeks in year 2, and every 12 weeks in year 3. Patients who lose their molecular remission may restart TKI medication and are monitored every 4 weeks in year 1, every 6 weeks in year 2, and every 12 weeks in year 3.
  Interventions: Procedure: Biospecimen Collection; Other: Drug Withdrawn; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tyrosine Kinase Inhibitor

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Drug Withdrawn — Stop taking TKI medication
  Other Names: discontinue (study treatment); Discontinued
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Tyrosine Kinase Inhibitor — Re-start TKI medication
  Other Names: Protein Tyrosine Kinase Inhibitors; PTK Inhibitors; TK Inhibitors

SUMMARY:
This phase II trial studies how stopping tyrosine kinase inhibitors will affect treatment-free remission in patients with chronic myeloid leukemia in chronic phase. When the level of disease is very low, it's called molecular remission. TKIs are a type of medication that help keep this level low. However, after being in molecular remission for a specific amount of time, it may not be necessary to take tyrosine kinase inhibitors. It is not yet known whether stopping tyrosine kinase inhibitors will help patients with chronic myeloid leukemia in chronic phase continue or re-achieve molecular remission.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 2-year treatment free remission (TFR) rate of children, adolescents, and young adults with chronic myeloid leukemia - chronic phase (CML-CP) following discontinuation tyrosine kinase inhibitor (TKI).

II. To estimate the re-induction rate and maintenance of molecular remission (BCR-ABL1 =< 0.1%) at 1 year after restarting TKI for children, adolescents, and young adults.

SECONDARY OBJECTIVE:

I. To describe clinical factors and laboratory correlates affecting the persistence of major molecular remission (MMR) and re-initiation of treatment after stopping TKI (e.g. patient demographics, duration and level of prior molecular remission, duration and type of TKI, clinical presentation at diagnosis and immune studies).

EXPLORATORY OBJECTIVES:

I. To describe change in height standard deviation score over time in patients who are able to discontinue their TKI.

II. To describe the long-term health outcomes including but not limited to gonadal function, endocrine function, and bone metabolism in patients who are able to discontinue TKI as well as those that need to restart TKIs.

III. To describe differences in patient-reported health status after stopping TKIs, including those who need to resume TKI after stopping.

IV. To describe the incidence and characteristics of TKI withdrawal syndrome in children.

V. To evaluate changes in neurocognitive outcomes of patients enrolled on this study using a patient-completed, performance-based, computerized measure of neuropsychological functioning and a parent-report/self-report questionnaire.

OUTLINE:

Patients stop taking TKI medication within 10 days after enrollment. Patients undergo peripheral blood collection to monitor loss of MMR every 4 weeks in year 1, every 6 weeks in year 2, and every 12 weeks in year 3. Patients who lose their molecular remission may restart TKI medication and are monitored every 4 weeks in year 1, every 6 weeks in year 2, and every 12 weeks in year 3.

After completion of study treatment, patients are followed up annually.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have been diagnosed with CML-CP at < 18 years of age.
* Patient must have histologic verification of CML-CP at original diagnosis
* Patient must be in molecular remission (MR) with a BCR-ABL1 level of =< 0.01% BCR-ABL1 as measured using the International Scale (IS) by RQ-PCR for >= 2 consecutive years at the time of enrollment

  * Please note: The lab evaluating disease status and molecular response for this study must be College of American Pathology (CAP) and/or Clinical Laboratory Improvement Amendments (CLIA) certified (United States [US] only), sites in other countries must be certified by their accredited authorities. All labs must use the International Scale guidelines with a sensitivity of detection assay =< 0.01% BCR-ABL1 and be able to report results in =< 2 weeks
* Patient must have received any TKI for a minimum of 3 consecutive years at time of enrollment
* Patient agrees to discontinue TKI therapy
* REGULATORY REQUIREMENTS
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met
* ELIGIBILITY FOR PATIENT-REPORTED OUTCOMES (PROs):
* Age >= 8 years at the time of enrollment
* Ability to understand English or Spanish
* Cognitive ability to complete instruments according to the primary team
* ELIGIBILITY FOR AAML18P1 NEUROCOGNITIVE STUDY:
* Patient must be 5 years or older at the time of enrollment
* English-, French- or Spanish-speaking
* No known history of neurodevelopmental disorder prior to diagnosis of CML (e.g., Down syndrome, Fragile X, William syndrome, mental retardation)
* No significant visual or motor impairment that would prevent computer use or recognition of visual test stimuli

Exclusion Criteria:

* Known T3151 mutation
* Additional clonal chromosomal abnormalities in Philadelphia chromosome (Ph) positive (+) cells at any time prior to enrollment that include "major route" abnormalities (second Ph, trisomy 8, isochromosome 17q, trisomy 19), complex karyotype or abnormalities of 3q26.2
* History of accelerated phase or blast crisis CML
* Female patients who are pregnant
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-free remission (TFR) | From date of TKI discontinuation to the date of the first event (molecular recurrence, hematologic relapse, cytogenetic relapse, re-initiation of TKI therapy, second malignant neoplasm, or death) or censoring, assessed up to 2 years
  The Kaplan Meier method will be used to estimate 2-year TFR along with a 95% confidence interval.
Major molecular remission (MMR/MR3) | Up to 1 year
  For patients re-initiating tyrosine kinase inhibitor (TKI) therapy, the cumulative incidence of major molecular remission will be calculated from the time of re-initiating TKI therapy treating deaths prior to achieving major molecular remission as competing events.

SECONDARY OUTCOMES:
Clinical factors and laboratory correlates affecting persistence of MMR | Up to 36 months
  Clinical factors and laboratory correlates (e.g. duration and level of prior molecular remission, risk score, duration and type of TKI, disease scoring system and immune studies etc.) affecting persistence of MMR and re-initiation of treatment after stopping TKI will be assessed by Cox proportional hazard regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Chaudhury, Principal Investigator — Children's Oncology Group
Locations (173):
- United States (157):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
- Australia (5):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico